CLINICAL TRIAL: NCT00003743
Title: Multicenter Observer-Blind Randomized Phase II Parallel Study Comparing Three Doses of Subcutaneous Interleukin 2 After Megatherapy and Peripheral Stem Cell Reinfusion in Stage 4 Neuroblastoma in Patients Over 1 Year of Age
Brief Title: Interleukin-2 in Treating Children With Stage IV Neuroblastoma Who Have Received Induction Therapy and Peripheral Stem Cell Transplantation
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: St. Anna Kinderkrebsforschung (Other)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Purpose: Treatment
Other Study IDs: CDR0000066861; STANNACH-INTERLEUKIN-2; EU-98056
Record Dates: First submitted 1999-11-01; First posted 2004-07-16 (Estimated); Last update posted 2013-09-17 (Estimated); Status verified 2007-05

CONDITIONS: Neuroblastoma
Keywords: disseminated neuroblastoma
MeSH Terms: conditions — Neuroblastoma | interventions — aldesleukin

INTERVENTIONS:
Biological: aldesleukin

SUMMARY:
RATIONALE: Interleukin-2 may stimulate a person's white blood cells to kill neuroblastoma cells.

PURPOSE: Phase II trial to study the effectiveness of interleukin-2 in treating children with stage IV neuroblastoma who have received induction therapy and peripheral stem cell transplantation.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the maximum dose that can be administered in an ambulatory setting among three dose regimens in children with stage IV neuroblastoma. II. Determine the highest tolerated level if a sustained increase in NK-cell number is observed. III. Determine the type, duration, and reversibility of side effects at the three dose levels. IV. Confirm the chosen dose level.

OUTLINE: This is a randomized, parallel, open label, multicenter study. Part I: Patients receive one of three doses of interleukin-2 (IL-2) subcutaneously beginning 20 to 40 days following autologous stem cell reinfusion. IL-2 is administered for 5 consecutive days every 14 days for up to 3 months, for a total of 6 courses. Cohorts of 5 patients are entered at each dose level of IL-2 until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose at which 3 or more patients experience dose limiting toxicity. Part II: Additional patients receive IL-2 at the dose level below the MTD. These patients are stratified according to prior therapy (melphalan plus megatherapy vs total body irradiation or meta-iodobenzylguanidine scan plus melphalan vs busulfan containing regimens). Patients are followed at 1 week.

PROJECTED ACCRUAL: Approximately 25 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically proven stage IV neuroblastoma At least stable disease after modern induction regimens and megatherapy followed by autologous stem cell reinfusion

PATIENT CHARACTERISTICS: Age: Over 1 Performance status: Lansky 80-100% Life expectancy: Not specified Hematopoietic: Lymphocyte count at least 500/mm3 Platelet count at least 30,000/mm3 Hemoglobin at least 8 g/dL (at least 1 week since transfusional support) Blood coagulation less than 25% above upper limit of normal (ULN) for age (WHO grade 0) Hepatic: Bilirubin less than 25% above ULN for age (WHO grade 0) Renal: Creatinine less than 25% above ULN for age (WHO grade 0) Cardiovascular: No significant history or current evidence of cardiovascular disease (e.g., uncontrolled hypertension, serious arrhythmias) Normal shortening fraction at cardiac ultrasonography Normal ECG Other: No evidence of active infections Normal chest x-ray Normal brain CT scan No other concurrent disease or second primary malignancy

PRIOR CONCURRENT THERAPY: Biologic therapy: See Disease Characteristics No other concurrent immunotherapy Chemotherapy: See Disease Characteristics No concurrent chemotherapy Endocrine therapy: No concurrent corticosteroids or other hormonal therapy Radiotherapy: No concurrent radiotherapy Surgery: Not specified Other: At least 30 days since prior investigational drugs or devices No concurrent investigational drugs, agents, or devices

Ages: 1 Year to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 25 (Estimated)
Dates: Start 1997-03

CONTACTS AND LOCATIONS:
Overall Officials: Ruth Ladenstein, MD, Study Chair — St. Anna Kinderkrebsforschung
Locations (1):
- St. Anna Children's Hospital, Vienna, Austria